CLINICAL TRIAL: NCT03440580
Title: BOOSTH: Promoting Physical Activity in Primary Schools in Combination With Serious Gaming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METC 172043
Record Dates: First submitted 2018-01-30; First posted 2018-02-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Physical Activity; Serious Game; Child Behavior; School Intervention
Keywords: physical activity; serious game; school intervention; children
MeSH Terms: conditions — Motor Activity; Child Behavior

STUDY DESIGN:
Intervention Model Description: The study design will be a randomized controlled trial regarding a physical activity intervention. A 1:1 randomization will be applied with intervention schools and matched control schools. The intervention school will recieve the BOOSTH intervention
Masking Description: Schools will be randomized into intervention or control schools. Randomization will be done by an independent researcher. After the randomization, the intervention school receives the BOOSTH intervention. The control school receives BOOSTH after the study is finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The intervention school will receive the BOOSTH intervention: Boosth activity tracker, Boosth sync app, Boosht game app
  Interventions: Device: BOOSTH
- control group (No Intervention): The control school will receive the standard curriculum. After the study is finished the children of the control school will receive the Boosth product

INTERVENTIONS:
Device: BOOSTH — BOOSTH as a serious game is used as a tool to motivate children to perform more PA. BOOSTH uses the combination of a smartphone game and a pedometer that assesses daily PA by measuring steps/day. The BOOSTH activity monitor is a wrist-worn activity monitor that is able to provide online feedback on the child's PA levels. Moreover, BOOSTH is a reward-based game as a child is given incentive to increase their PA level, in order to acquire activity points which later can be used to unlock levels and progress in the BOOSTH game.
  Arms: Intervention

SUMMARY:
Physical inactivity is considered to be one of the ten principal risk factors for death worldwide. Children need to perform one hour of daily moderate-to-vigorous intensity physical activity whereof at least twice a week these activities are of vigorous intensity. In 2010, the percentage of 4-11 year-old normoactive Dutch children was approximately 20%.Previous interventions that aimed to increase childhood physical activity produced small to negligible effects. One possible explanation is that individuals were not intrinsically motivated towards physical activity during the intervention period. Children spend a substantial amount of their time behind a game consule. There are a number of applications that motivate increase in physical activity in a fun way through engaging individuals in games that mix real and computing worlds. These games became known as serious games. In this study we want to investigate if the incorporation of a serious game BOOSTH in combination with an activity tracker and battle to stimulate physical activity behaviour in primary school children (grades 5th to 7th).

DETAILED DESCRIPTION:
The study design will be a randomized controlled trial regarding a physical activity intervention. A 1:1 randomization will be applied with intervention schools and matched control schools. The intervention school will recieve the BOOSTH intervention. The intervention duration is 6 months. Measurements will be performed at baseline and 3, 6 and 12 months after the start.

The investigational treatment is the BOOSTH physical activity intervention. Children in the intervention school will start with the BOOSTH intervention on top of the regular PE lessons. The child will receive the BOOSTH activity tracker. The child (under supervision of the teacher) needs to download the BOOSTH sync app and the BOOSTH game app. Therefore it is important that the school works with a device with Bluetooth. We will create a login account for each child. After installing the apps, the activity tracker measures step counts, which are translated into activity points. These activity points will be used to unlock levels in the BOOSTH game app. The child synchronizes their activity points, with Bluetooth connection, in the BOOSTH sync app and immediately the child can open the BOOSTH game app to play a level in the game. The child needs seven green lights (corresponding to 30 minutes of performed physical activity) to unlock a level in the game. The first four levels are for free, to gain the interests of the child, but thereafter the child needs to be physically active to unlock the rest of the levels in the game.

ELIGIBILITY:
Inclusion criteria:

* The school needs to be located in the Limburg- region of the Netherlands.
* At least 25 students enrolled in grades 5, 6 and 7
* The school works with a technological device with Bluetooth option to synchronize activity points
* Boys and girls, in 5th to 7th grade
* Informed consent signed by both parents and children aged 12 years and older.

Exlusion criteria

* Children who are wheelchair dependent.
* The school has plans to merge with another school or plans to relocate in the upcoming year.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 713 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
moderate to vigorous physical activity (min/day) | up to twelve months
  change in moderate to vigorous physical activity (min/day) as measured with accelerometry

SECONDARY OUTCOMES:
change in step count | up to twelve months
  step count as measured with the Boosth activity tracker
change in physical activity behaviour | up to twelve months
  subjectively measured physical activity behaviour with BAECKE questionnaire. BAECKE (for children) will be used to assess the amount of habitual PA ranging from 1 (lowest activity) to 5 (highest activity). Physical activity at school, during leisure time and organized sports will be asked.
BMI-z score | up to twelve months
  change in BMI- z score. BMI is calculated as weight (kilograms) divided by height (meters) squared. for children the BMI threshold of obesity varies with age and sex.
motivation towards physical activity | up to twelve months (measurement at baseline,3-, 6- and 12 months)
  motivation towards physical activity as measured with BREQ questionnaire. The BREQ2 is a self-administered questionnaire about a motivation continuum towards PA. The BREQ2 measures external, introjected, identified, integrated and intrinsic forms of motivation of PA behavior. The questionnaire consists of 19 thesis's on a 5-point Likert scale, providing subscores for all forms of regulation. The BREQ2 is a self-administered questionnaire about a motivation continuum towards PA. The BREQ2 measures external, introjected, identified, integrated and intrinsic forms of motivation of PA behavior. The questionnaire consists of 19 thesis's on a 5-point Likert scale, providing subscores for all forms of regulation.
screen-time | up to twelve months (measurement at baseline,3-, 6- and 12 months)
  screen- time as measured with questionnaire. Self-reported screen time will be reported separately for weekday and weekend day assessed with the following questions: 'How many hours a day during the last 4 weeks you watched TV on a normal weekday/weekend?' and 'How many hours a day during the last 4 weeks have you played console games or used a computer for your free time activities on a normal weekday/weekend? Possible responses are: 'not at all', '0.5 hours per day', 'one hour per day', '2 hours per day', '2.5 hours per day', '3 hours per day', '3.5 hours per day', '4 hours or more per day'. Total screen time was calculated by summing minutes spent in TV watching and computer use.
Quality of life (Kidscreen) | up to twelve months (measurement at baseline,3-, 6- and 12 months)
  Quality of life as measured with Kidscreen. The Kidsreen instruments assess children's and adolescents' subjective health and well-being. They were developed as self-report measures applicable for healthy and chronically ill children and adolescents aged from 8 to 18 years. The Kidsscreen-27 version provides a global health related quality of life score and consists of 27 questions.Higher scores represent a better quality of life
Quality of life (PedsQL) | up to twelve months (measurement at baseline,3-, 6- and 12 months)
  Quality of life as measured with PedsQL questionnaire. The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. The 4 Multidimensional Scales are: physical functioning, emotional functioning, social functioning and school functioning. Summary scores will be calculated for total scale score, physical health summary score and psychosocial health summary score.
Cardiovascular alterations (Pulse Wave Velocity) | up to twelve months (measurement at baseline and 12 months)
  pulse wave velocity (PWV). will be measured using a SphygmoCor (CPV) device. Carotidfemoral (cf) as well as -radial (cr) PWV will be measured. Measurement of cr PWV in addition to cf PWV is no extra burden to the subjects and will take only a few extra minutes. Obtained waveforms are processed with dedicated software (SphygmoCor version 7, AtCor).
Blood pressure | up to twelve months (measurement at baseline and 12 months)
  blood pressure. Systolic and diastolic blood pressure will be measured using a validated automatic device on the right arm after 5-10 minutes rest in a resting position. The measurement is taken three times with a 1 minute rest between, and the reading is recorded to the nearest 1 mmHg. A mean value of these three readings is used
Cardiovascular alterations (retinal image) | up to twelve months (measurement at baseline and 12 months)
  Retinal image. Children are seated with the head resting on a chinrest, looking directly into the camera (Topcon TRC-NW-300, Topcon Corporation, Tokyo, Japan). The fundus camera will focus on and take a picture of the retina. The total procedure will take about 2 minutes. Images will be digitised and analysed to calculate the arteriovenous ratio (AVratio) with the appropriate software (Generalized Dual-Bootstrap Iterative Closest Point (GDB-ICP)) that is able to automatically initialise and individually match vascular landmarks. In addition, the software will be used to measure the diameter of the four largest retinal arterioles and venules
Aerobic fitness | up to twelve months (measurement at baseline and 12 months)
  aerobic fitness as measured with the 20m shuttle run test

OTHER OUTCOMES:
Comprehensive General Parenting Questionnaire | up to twelve months (measurement at baseline and 6 months)
  Parenting style as measured with CGPQ. The 85 item Comprehensive General Parenting Questionnaire (CGPQ) will be used to assess general parenting on a five - factor parenting model. This questionnaire is validated with Dutch parents questionnaire.
parenting practices questionnaire | up to twelve months (measurement at baseline and 6 months)
  Parenting style as measured with parenting practices questionnaire. The physical activity parenting practice questionnaire assess parents practice style regarding physical activity and sedentary behavior. The questionnaire consists of 5 questions on a 5point scale.
Process evaluation | up to 6 months (measurement at 3- and 6 months)
  Process evaluation Semi- structured focus groups will be caried out with teachers from the intervention schools. The interview covers all aspects of the intervention, including the measurements, introduction lesson of Boosth, the intervention and the follow up. Interviews will be recorded. Booking logs: will be used to assess intervention reach and dose. Evaluation questionnaire: children and their parents will fill in an evaluation questionnaire about the use of BOOSTH. Teachers will fill in an evaluation questionnaire about the methods and implementation about the BOOSTH intervention. Teachers of the control school will fill in an questionnaire to find out whether any unplanned intervention may contaminated the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, Dr, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Velde GT, Plasqui G, Willeboordse M, Winkens B, Vreugdenhil A. Associations between physical activity, sedentary time and cardiovascular risk factors among Dutch children. PLoS One. 2021 Aug 27;16(8):e0256448. doi: 10.1371/journal.pone.0256448. eCollection 2021. PMID 34449807
- [Derived] Ten Velde G, Plasqui G, Willeboordse M, Winkens B, Vreugdenhil A. Feasibility and Effect of the Exergame BOOSTH Introduced to Improve Physical Activity and Health in Children: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 11;9(12):e24035. doi: 10.2196/24035. PMID 33306031